CLINICAL TRIAL: NCT00174291
Title: Prevention of Retarded Growth by Early Treatment With Recombinant Human Growth Factor Genotonorm (Registered) in Children With Systemic Forms of Chronic Juvenile Arthritis Receiving Long-term Corticosteroid Therapy. Extension of the Study Beyond Three Years
Brief Title: Prevention of Growth Retardation by Early Treatment With Growth Hormone (GH) in Children With CJA Treated by Corticosteroid Therapy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 307-MET-9002-052; A6281024
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Results first posted 2012-12-04 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-10

CONDITIONS: Endocrine System Diseases
MeSH Terms: conditions — Endocrine System Diseases | interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Somatropin (Experimental)
  Interventions: Drug: Somatropin

INTERVENTIONS:
Drug: Somatropin — Liquid, daily to final height Maximum Dosage: 50 µg/kg/day

SUMMARY:
* To evaluate the effect of increasing the growth hormone dose on the statural response
* To assess the value of early treatment during the course of arthritic disease by comparing the height acquired in the medium term by children in the two groups: treated from the start, or 1 year to 15 months after the diagnosis of CJA, or treated for 4 years after the diagnosis

DETAILED DESCRIPTION:
This trial terminated on 10-Jun-2011 due to prolonged issues with drug accountability and data collection discrepancies. The decision to terminate was not based on any safety concerns.

ELIGIBILITY:
Inclusion Criteria:

* This study will be proposed to all patients previously included in study CTN 97-8129-016

Exclusion Criteria:

* Discontinuation of corticosteroid therapy for more than a year during study CTN 97-8129-016
* Patients withdrawing from the study prematurely

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2002-03; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Paris, France

REFERENCES:
- [Derived] David H, Aupiais C, Louveau B, Quartier P, Jacqz-Aigrain E, Carel JC, Simon D. Growth Outcomes After GH Therapy of Patients Given Long-Term Corticosteroids for Juvenile Idiopathic Arthritis. J Clin Endocrinol Metab. 2017 Dec 1;102(12):4578-4587. doi: 10.1210/jc.2017-01455. PMID 29029101
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=307-MET-9002-052&StudyName=Prevention%20of%20Growth%20Retardation%20by%20Early%20Treatment%20with%20Growth%20Hormone%20%28GH%29%20in%20Children%20with%20CJA%20Treated%20by%20Corticosteroid%20Th

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants included in previous study CTN 97-8129-016 were eligible for this study.
Groups:
- Somatropin (With Previous Somatropin Exposure): Participants who received low dose of somatropin (Genotonorm) for 3 years during previous study CTN 97-8129-016, received somatropin (Genotonorm) up to 0.6 milligram per kilogram per week (mg/kg/week), equivalent to 1.8 international units/kg/week (IU/kg/week), divided in 7 daily doses subcutaneously initially for first 3 years and then somatropin (Genotonorm) 0.46 mg/kg/week, equivalent to 1.4 IU/kg/week, divided in 7 daily doses subcutaneously until the additional study drug dose evaluation visit and thereafter received somatropin (Genotonorm) 50 microgram/kg/day (mcg/kg/day), equivalent to 0.35 mg/kg/week or 1.05 IU/kg/week, subcutaneously until the final height was reached or up to Year 8.5. Final height was confirmed to have been achieved if the growth velocity was less than or equal to 1.5 centimeter (cm) per year during the preceding 12 months and bone age was greater than or equal to 17 years for boys and 15 years for girls.
- Somatropin (Without Previous Somatropin Exposure): Participants who received matching placebo for 3 years during previous study CTN 97-8129-016, received somatropin (Genotonorm) up to 0.6 mg/kg/week, equivalent to 1.8 IU/kg/week, divided in 7 daily doses subcutaneously initially for first 3 years and then somatropin (Genotonorm) 0.46 mg/kg/week, equivalent to 1.4 IU/kg/week, divided in 7 daily doses subcutaneously until the additional study drug dose evaluation visit and thereafter received somatropin (Genotonorm) 50 mcg/kg/day, equivalent to 0.35 mg/kg/week or 1.05 IU/kg/week, subcutaneously until the final height was reached or up to Year 8.5. Final height was confirmed to have been achieved if the growth velocity was less than or equal to 1.5 cm per year during the preceding 12 months and bone age was greater than or equal to 17 years for boys and 15 years for girls.
Period: Overall Study
Arm/Group | Somatropin (With Previous Somatropin Exposure) | Somatropin (Without Previous Somatropin Exposure)
Started | 11 | 10
Completed | 6 | 4
Not Completed | 5 | 6
Not completed — Lost to Follow-up | 1 | 1
Not completed — Protocol Violation | 0 | 2
Not completed — Study terminated by sponsor | 1 | 0
Not completed — Withdrawal by Subject | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Somatropin (With Previous Somatropin Exposure) | Somatropin (Without Previous Somatropin Exposure) | Total
Number analyzed (Participants) | 11 | 10 | 21
Age Continuous [Mean (Standard Deviation); unit: years] | 8.3 (2.6) | 8.5 (3.3) | 8.4 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Annual Rate of Growth Standard Deviation Score (SDS) at Year 3
Description: Annual rate of growth SDS was obtained by measuring the annual growth rate, subtracting chronological age- and gender-appropriate mean annual growth rate and dividing the result by standard deviation of that mean (as obtained from chronological age- and gender-specific population reference data). SDS indicated how many standard deviations higher (in case of positive SDS) or lower (in case of negative SDS) participant's value was relative to the mean of the reference population.
Time Frame: Baseline, Year 3
Population: Full Analysis Set (FAS) included all participants who received at least 1 dose of study treatment and had at least 1 post-baseline height measurement. Here, N (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Median (Full Range); unit: SDS
Arm/Group | Somatropin (With Previous Somatropin Exposure) | Somatropin (Without Previous Somatropin Exposure)
Number analyzed (Participants) | 6 | 9
SDS
  Baseline | -0.21 [-3.0 to 4.5] | -2.96 [-6.4 to 1.5]
  Change at Year 3 | 1.34 [-3.6 to 6.2] | 3.52 [-5.1 to 11.2]

2. Primary Outcome: Change From Baseline in Annual Rate of Growth Standard Deviation Score (SDS) at Final Height
Description: as for outcome 1
Time Frame: Baseline, final height (assessed up to Year 9.5)
Population: Data was not analyzed because of change in planned analysis after early termination of the study.
Arm/Group | Somatropin (With Previous Somatropin Exposure) | Somatropin (Without Previous Somatropin Exposure)
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Change From Baseline in Height Standard Deviation Score (SDS) at Year 3
Description: Height was measured using a wall mounted device (example, Harpenden stadiometer). Height SDS was obtained by measuring the height, subtracting chronological age- and gender-appropriate mean height and dividing the result by standard deviation of that mean (as obtained from chronological age- and gender-specific population reference data). SDS indicated how many standard deviations higher (in case of positive SDS) or lower (in case of negative SDS) participant's value was relative to the mean of the reference population.
Time Frame: Baseline, Year 3
Population: FAS included all participants who received at least 1 dose of study treatment and had at least 1 post-baseline height measurement. Here, N (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Median (Full Range); unit: SDS
Arm/Group | Somatropin (With Previous Somatropin Exposure) | Somatropin (Without Previous Somatropin Exposure)
Number analyzed (Participants) | 6 | 9
SDS
  Baseline | -0.61 [-3.7 to 1.4] | -2.34 [-4.8 to -1.4]
  Change at Year 3 | 0.73 [-2.4 to 2.6] | 1.21 [-0.7 to 2.4]

4. Primary Outcome: Change From Baseline in Height Standard Deviation Score (SDS) at Final Height
Description: as for outcome 3
Time Frame: Baseline, final height (assessed up to Year 9.5)
Population: as for outcome 3
Measure: Median (Full Range); unit: SDS
Arm/Group | Somatropin (With Previous Somatropin Exposure) | Somatropin (Without Previous Somatropin Exposure)
Number analyzed (Participants) | 3 | 2
SDS
  Baseline | 0.96 [-3.7 to 2.3] | -0.94 [-1.4 to -0.5]
  Change at Final Height | -0.43 [-0.8 to 0.5] | 0.08 [-0.7 to 0.9]

5. Primary Outcome: Change From Baseline in Predicted Height Standard Deviation Score (SDS) at Year 3
Description: Predicted height was calculated according to Greulich and Pyle using Bayley Pinneau method. Predicted height SDS was obtained by calculating the predicted height, subtracting chronological age- and gender-appropriate mean predicted height and dividing the result by standard deviation of that mean (as obtained from chronological age- and gender-specific population reference data). SDS indicated how many standard deviations higher (in case of positive SDS) or lower (in case of negative SDS) participant's value was relative to the mean of the reference population.
Time Frame: Baseline, Year 3
Population: as for outcome 3
Measure: Median (Full Range); unit: SDS
Arm/Group | Somatropin (With Previous Somatropin Exposure) | Somatropin (Without Previous Somatropin Exposure)
Number analyzed (Participants) | 4 | 3
SDS
  Baseline | -0.76 [-1.8 to 0.7] | -2.43 [-2.6 to -1.6]
  Change at Year 3 | 0.68 [-2.6 to 2.0] | 1.63 [0.1 to 2.3]

6. Primary Outcome: Change From Baseline in Predicted Height Standard Deviation Score (SDS) at Final Height
Description: as for outcome 5
Time Frame: Baseline, final height (assessed up to Year 9.5)
Population: as for outcome 3
Measure: Median (Full Range); unit: SDS
Arm/Group | Somatropin (With Previous Somatropin Exposure) | Somatropin (Without Previous Somatropin Exposure)
Number analyzed (Participants) | 2 | 2
SDS
  Baseline | -0.84 [-1.8 to 0.1] | -1.74 [-2.4 to -1.1]
  Change at Final Height | -0.67 [-2.4 to 1.0] | 0.71 [0.1 to 1.3]

7. Secondary Outcome: Change From Baseline in Insulin-like Growth Factor-1 (IGF-1) Concentration at Year 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5, 8, 8.5 and 9
Time Frame: Baseline, Year 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5, 8, 8.5, 9
Population: FAS included all participants who received at least 1 dose of study treatment and had at least 1 post-baseline height measurement. Here, 'n' signifies those participants who were evaluable for this measure at given time points for each group respectively.
Measure: Median (Full Range); unit: milligram per deciliter (mg/dL)
Arm/Group | Somatropin (With Previous Somatropin Exposure) | Somatropin (Without Previous Somatropin Exposure)
Number analyzed (Participants) | 11 | 10
milligram per deciliter (mg/dL)
  Baseline (n = 11, 10) | 0.0361 [0.0181 to 0.0868] | 0.0165 [0.0075 to 0.0517]
  Change at Year 0.5 (n = 9, 10) | 0.0017 [-0.0256 to 0.0681] | 0.0255 [-0.0145 to 0.0390]
  Change at Year 1 (n = 11, 10) | 0.0093 [-0.0358 to 0.0488] | 0.0329 [-0.0061 to 0.0531]
  Change at Year 1.5 (n = 11, 9) | 0.0066 [-0.0194 to 0.0599] | 0.0406 [-0.0035 to 0.0754]
  Change at Year 2 (n = 10, 9) | 0.0221 [-0.0292 to 0.0534] | 0.0223 [0.0055 to 0.0673]
  Change at Year 2.5 (n = 8, 8) | 0.0201 [-0.0237 to 0.0470] | 0.0366 [-0.0109 to 0.0558]
  Change at Year 3 (n = 7, 9) | 0.0130 [-0.0049 to 0.0648] | 0.0445 [-0.0060 to 0.0557]
  Change at Year 3.5 (n = 7, 7) | 0.0100 [-0.0022 to 0.0436] | 0.0396 [0.0014 to 0.0707]
  Change at Year 4 (n = 6, 7) | 0.0212 [-0.0014 to 0.0485] | 0.0453 [0.0175 to 0.0646]
  Change at Year 4.5 (n = 5, 6) | 0.0142 [0.0042 to 0.0303] | 0.0431 [0.0080 to 0.1233]
  Change at Year 5 (n = 5, 7) | 0.0236 [0.0164 to 0.0530] | 0.0369 [0.0258 to 0.0902]
  Change at Year 5.5 (n = 4, 5) | 0.0186 [0.0119 to 0.0356] | 0.0448 [0.0258 to 0.0965]
  Change at Year 6 (n = 4, 5) | 0.0256 [0.0000 to 0.0434] | 0.0454 [0.0155 to 0.0718]
  Change at Year 6.5 (n = 2, 5) | 0.0195 [0.0125 to 0.0264] | 0.0593 [0.0512 to 0.0766]
  Change at Year 7 (n = 1, 5) | 0.0254 [0.0254 to 0.0254] | 0.0424 [0.0393 to 0.0766]
  Change at Year 7.5 (n = 0, 3) | NA [NA to NA] — Data were not analyzed since none of the participants were available in this group at given time point. | 0.0529 [0.0527 to 0.0599]
  Change at Year 8 (n = 0, 2) | NA [NA to NA] — Data were not analyzed since none of the participants were available in this group at given time point. | 0.0576 [0.0468 to 0.0683]
  Change at Year 8.5 (n = 0, 1) | NA [NA to NA] — Data were not analyzed since none of the participants were available in this group at given time point. | 0.0280 [0.0280 to 0.0280]
  Change at Year 9 (n = 2, 1) | 0.0363 [0.0159 to 0.0567] | 0.0403 [0.0403 to 0.0403]

8. Secondary Outcome: Change From Baseline in Insulin-like Growth Factor Binding Protein 3 (IGFBP3) Concentration at Year 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5, 8, 8.5 and 9
Time Frame: Baseline, Year 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5, 8, 8.5, 9
Population: Data were collected and reported in individual participant listing but not statistically summarized due to early termination of the study.
Arm/Group | Somatropin (With Previous Somatropin Exposure) | Somatropin (Without Previous Somatropin Exposure)
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Change From Baseline in Lean Mass and Fat Mass at Year 1, 2, 3, 4, 5, 6, 7, 8 and 9
Description: Lean mass and fat mass: measurements of body composition assessed using Dual Energy X-ray Absorptiometry (DEXA) scan.
Time Frame: Baseline, Year 1, 2, 3, 4, 5, 6, 7, 8, 9
Population: as for outcome 8
Arm/Group | Somatropin (With Previous Somatropin Exposure) | Somatropin (Without Previous Somatropin Exposure)
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Change From Baseline in Bone Mineralization at Year 1, 2, 3, 4, 5, 6, 7, 8 and 9
Description: Bone mineralization, an estimate of the amount of mineral (such as calcium) in the bone, was assessed using DEXA scan.
Time Frame: Baseline, Year 1, 2, 3, 4, 5, 6, 7, 8, 9
Population: as for outcome 7
Measure: Median (Full Range); unit: grams
Arm/Group | Somatropin (With Previous Somatropin Exposure) | Somatropin (Without Previous Somatropin Exposure)
Number analyzed (Participants) | 11 | 10
grams
  Baseline (n = 11, 10) | 643.00 [454.0 to 998.0] | 565.40 [136.0 to 1305.0]
  Change at Year 1 (n = 11, 10) | 118.40 [-792.7 to 459.6] | 104.67 [9.0 to 340.0]
  Change at Year 2 (n = 10, 9) | 231.30 [-47.5 to 774.4] | 272.70 [63.0 to 590.0]
  Change at Year 3 (n = 7, 8) | 403.80 [25.0 to 862.5] | 375.27 [106.0 to 1084.9]
  Change at Year 4 (n = 4, 3) | 903.20 [277.1 to 1448.1] | 518.70 [450.8 to 1047.9]
  Change at Year 5 (n = 4, 7) | 938.30 [591.8 to 1787.6] | 829.00 [421.7 to 1245.8]
  Change at Year 6 (n = 4, 5) | 998.05 [371.4 to 1984.2] | 818.40 [112.5 to 1105.5]
  Change at Year 7 (n = 1, 5) | 1408.50 [1408.5 to 1408.5] | 1206.10 [739.6 to 1437.3]
  Change at Year 8 (n = 0, 2) | NA [NA to NA] — Data were not analyzed since none of the participants were available in this group at given time point. | 1376.05 [1351.7 to 1400.4]
  Change at Year 9 (n = 2, 1) | 1210.15 [898.6 to 1521.7] | 1376.30 [1376.3 to 1376.3]

11. Secondary Outcome: Change From Baseline in Weight Standard Deviation Score (SDS) at Year 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5, 8, 8.5 and 9
Description: Body weight was measured using a balance scale. Weight SDS was obtained by measuring the weight, subtracting age- and gender- appropriate mean weight and dividing the result by standard deviation of that mean (as obtained from age- and gender-specific population reference data). SDS indicated how many standard deviations higher (in case of positive SDS) or lower (in case of negative SDS) participant's value was relative to the mean of the reference population.
Time Frame: Baseline, Year 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5, 8, 8.5, 9
Population: as for outcome 7
Measure: Median (Full Range); unit: SDS
Arm/Group | Somatropin (With Previous Somatropin Exposure) | Somatropin (Without Previous Somatropin Exposure)
Number analyzed (Participants) | 11 | 10
SDS
  Baseline (n = 11, 10) | 0.04 [-5.4 to 5.0] | -2.06 [-4.0 to 2.6]
  Change at Year 0.5 (n = 9, 10) | 0.06 [-0.8 to 1.2] | 0.25 [-0.7 to 0.4]
  Change at Year 1 (n = 11, 10) | 0.25 [-1.1 to 0.9] | 0.31 [-0.1 to 1.5]
  Change at Year 1.5 (n = 11, 9) | 0.34 [-1.6 to 2.3] | 0.62 [-0.3 to 2.3]
  Change at Year 2 (n = 10, 9) | 0.46 [-1.1 to 2.2] | 1.23 [-0.2 to 2.7]
  Change at Year 2.5 (n = 8, 8) | 0.77 [-1.1 to 2.6] | 1.51 [-0.9 to 3.2]
  Change at Year 3 (n = 7, 9) | 0.61 [-1.2 to 2.7] | 1.48 [-1.9 to 3.7]
  Change at Year 3.5 (n = 7, 7) | 0.78 [-1.3 to 3.0] | 1.56 [-1.9 to 3.7]
  Change at Year 4 (n = 6, 7) | 0.58 [-1.0 to 2.4] | 1.96 [-2.3 to 3.8]
  Change at Year 4.5 (n = 5, 6) | 1.46 [-0.4 to 2.7] | 1.78 [-2.7 to 4.1]
  Change at Year 5 (n = 5, 7) | 2.06 [0.1 to 2.8] | 2.08 [-3.0 to 3.9]
  Change at Year 5.5 (n = 3, 5) | 2.10 [1.7 to 2.6] | 3.25 [1.0 to 3.8]
  Change at Year 6 (n = 3, 5) | 1.89 [1.8 to 2.2] | 2.95 [1.2 to 4.4]
  Change at Year 6.5 (n = 2, 5) | 2.03 [1.9 to 2.2] | 3.30 [0.8 to 5.0]
  Change at Year 7 (n = 1, 5) | 1.7 [1.7 to 1.7] | 2.91 [0.2 to 5.2]
  Change at Year 7.5 (n = 0, 3) | NA [NA to NA] — Data were not analyzed since none of the participants were available in this group at given time point. | 1.49 [0.3 to 3.1]
  Change at Year 8 (n = 0, 2) | NA [NA to NA] — Data were not analyzed since none of the participants were available in this group at given time point. | 1.06 [0.5 to 1.6]
  Change at Year 8.5 (n = 0, 1) | NA [NA to NA] — Data were not analyzed since none of the participants were available in this group at given time point. | 0.7 [0.7 to 0.7]
  Change at Year 9 (n = 1, 1) | 2.0 [2.0 to 2.0] | 1.4 [1.4 to 1.4]

12. Secondary Outcome: Change From Baseline in Corticosteroid Dose at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5, 8, 8.5 and 9
Time Frame: Baseline, Year 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5, 8, 8.5, 9
Population: as for outcome 7
Measure: Median (Full Range); unit: mg
Arm/Group | Somatropin (With Previous Somatropin Exposure) | Somatropin (Without Previous Somatropin Exposure)
Number analyzed (Participants) | 11 | 10
mg
  Baseline (n = 11, 10) | 7.50 [1.0 to 40.0] | 4.75 [2.0 to 13.5]
  Change at Year 0.5 (n = 9, 10) | 0.00 [-11.0 to 0.0] | 0.00 [-2.5 to 4.8]
  Change at Year 1 (n = 11, 9) | 0.00 [-15.0 to 20.3] | -0.67 [-8.5 to 36.0]
  Change at Year 1.5 (n = 11, 8) | 0.00 [-17.0 to 7.5] | 0.50 [-5.0 to 8.8]
  Change at Year 2 (n = 10, 8) | 0.00 [-19.0 to 10.6] | -0.50 [-6.3 to 11.9]
  Change at Year 2.5 (n = 8, 7) | 0.04 [-28.0 to 7.5] | 1.83 [-7.8 to 11.9]
  Change at Year 3 (n = 7, 7) | 0.00 [-34.2 to 1.0] | 1.75 [-9.5 to 19.4]
  Change at Year 3.5 (n = 7, 6) | -0.75 [-36.0 to 2.9] | 1.83 [-10.3 to 12.5]
  Change at Year 4 (n = 6, 7) | -1.88 [-4.5 to 0.0] | 0.25 [-10.0 to 9.7]
  Change at Year 4.5 (n = 5, 6) | -3.40 [-10.0 to 0.0] | 0.23 [-9.0 to 215.4]
  Change at Year 5 (n = 5, 7) | -3.50 [-10.0 to -0.6] | -2.00 [-9.5 to 15.0]
  Change at Year 5.5 (n = 4, 5) | -1.83 [-4.5 to 486.5] | 0.25 [-9.5 to 18.3]
  Change at Year 6 (n = 4, 5) | -1.83 [-5.5 to 9.0] | -1.00 [-11.0 to 10.6]
  Change at Year 6.5 (n = 2, 5) | -2.46 [-3.7 to -1.3] | -1.00 [-11.0 to 3.0]
  Change at Year 7 (n = 1, 5) | -2.50 [-2.5 to -2.5] | -1.00 [-11.0 to 2.0]
  Change at Year 7.5 (n = 0, 3) | NA [NA to NA] — Data were not analyzed since none of the participants were available in this group at given time point. | -7.00 [-12.0 to 0.5]
  Change at Year 8 (n = 0, 2) | NA [NA to NA] — Data were not analyzed since none of the participants were available in this group at given time point. | -3.25 [-7.0 to 5.0]
  Change at Year 8.5 (n = 0, 1) | NA [NA to NA] — Data were not analyzed since none of the participants were available in this group at given time point. | 0.50 [0.5 to 0.5]
  Change at Year 9 (n = 2, 1) | -3.00 [-3.5 to -2.5] | -7.00 [-7.0 to -7.0]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Somatropin (With Previous Somatropin Exposure) | Somatropin (Without Previous Somatropin Exposure)
Serious Adverse Events (participants affected / at risk) | 6/11 | 2/10
Other Adverse Events (participants affected / at risk) | 11/11 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Somatropin (With Previous Somatropin Exposure) (N=11) | Somatropin (Without Previous Somatropin Exposure) (N=10)
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1
Hip dysplasia (Congenital, familial and genetic disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0
Leishmaniasis (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 0 | 1
Relapsing fever (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1
Juvenile arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Osteochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Histiocytosis haematophagic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Glomerulonephritis (Renal and urinary disorders) | 1 | 0
Nephrotic syndrome (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lipoatrophy (Skin and subcutaneous tissue disorders) | 1 | 0
Gastrostomy closure (Surgical and medical procedures) | 1 | 0
Hip arthroplasty (Surgical and medical procedures) | 1 | 0
Tooth extraction (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Somatropin (With Previous Somatropin Exposure) (N=11) | Somatropin (Without Previous Somatropin Exposure) (N=10)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Blood disorder (Blood and lymphatic system disorders) | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 1
Congenital scoliosis (Congenital, familial and genetic disorders) | 1 | 0
Hyperparathyroidism (Endocrine disorders) | 0 | 1
Cataract (Eye disorders) | 2 | 0
Conjunctivitis (Eye disorders) | 0 | 1
Visual acuity reduced (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Functional gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 2
Sigmoiditis (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 0 | 2
Ill-defined disorder (General disorders) | 2 | 1
Inflammation (General disorders) | 0 | 1
Influenza like illness (General disorders) | 1 | 0
Injection site haemorrhage (General disorders) | 0 | 1
Nodule (General disorders) | 0 | 1
Oedema (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 1
Hepatomegaly (Hepatobiliary disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 3
Ear infection (Infections and infestations) | 1 | 2
Gastroenteritis (Infections and infestations) | 2 | 1
Herpes simplex (Infections and infestations) | 0 | 1
Herpes virus infection (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 2
Infectious mononucleosis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Laryngitis (Infections and infestations) | 1 | 1
Nail candida (Infections and infestations) | 0 | 2
Nasopharyngitis (Infections and infestations) | 2 | 2
Oral herpes (Infections and infestations) | 1 | 0
Otitis externa (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 1
Tracheitis (Infections and infestations) | 0 | 1
Varicella (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 2 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 2
Procedural vomiting (Injury, poisoning and procedural complications) | 0 | 1
Blood corticotrophin decreased (Investigations) | 2 | 0
Blood glucose decreased (Investigations) | 1 | 0
Blood urine present (Investigations) | 0 | 1
Glucose tolerance test (Investigations) | 1 | 0
Glycosylated haemoglobin increased (Investigations) | 0 | 2
Insulin-like growth factor increased (Investigations) | 8 | 6
Weight decreased (Investigations) | 1 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 5 | 0
Hyperinsulinaemia (Metabolism and nutrition disorders) | 0 | 1
Insulin resistance (Metabolism and nutrition disorders) | 6 | 5
Amyotrophy (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 2 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Juvenile arthritis (Musculoskeletal and connective tissue disorders) | 4 | 4
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Hyporeflexia (Nervous system disorders) | 1 | 0
Hypotonia (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Visual field defect (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Nightmare (Psychiatric disorders) | 1 | 0
Sleep disorder (Psychiatric disorders) | 1 | 2
Enuresis (Renal and urinary disorders) | 0 | 2
Hypercalciuria (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 2 | 0
Gynaecomastia (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acanthosis nigricans (Skin and subcutaneous tissue disorders) | 1 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Lividity (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Skin atrophy (Skin and subcutaneous tissue disorders) | 1 | 0
Walking disability (Social circumstances) | 1 | 0
Knee operation (Surgical and medical procedures) | 0 | 1
Hypertension (Vascular disorders) | 1 | 1
Poor peripheral circulation (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Data for bone mineral density (BMD), bone mineral content (BMC) and IGFBP3 were not analyzed because of change in planned analysis after the study was prematurely terminated due to Good Clinical Practice (GCP) non-compliance issues.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.